CLINICAL TRIAL: NCT02574442
Title: Pilot Study of the Hand-held In Vivo Confocal Microscopy Probe for Detection of Cervical Intraepithelial Neoplasia
Brief Title: Pilot Study In Vivo Confocal Microscopy Probe for Cervical Precancer
Acronym: Confocal
Status: Terminated | Type: Observational
Why Stopped: Funding has run out
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BCCR - H15-01726; P01CA082710 (NIH); H15-01726 (Other: UBC BCCA REB)
Record Dates: First submitted 2015-09-01; First posted 2015-10-12 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Precancerous Condition; Cervical Cancer
Keywords: cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3; adenocarcinoma in situ
MeSH Terms: conditions — Precancerous Conditions; Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Adenocarcinoma in Situ

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cervical biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Initial Colposcopy Visit: Women with a scheduled colposcopy and biopsy appointment at the Women's Clinic at Vancouver General Hospital
  Interventions: Device: In Vivo Confocal Microscopy Probe

INTERVENTIONS:
Device: In Vivo Confocal Microscopy Probe — Participants will have 2 areas on their cervical imaged by the confocal probe.

SUMMARY:
The goal of this proposal is to determine whether a hand-held confocal microscopy probe may perform better than standard methods in detecting cancer or pre-cancerous abnormalities of the cervix. The confocal probe will provide invivo histopathology-like images of cell morphology and three-dimensional tissue architecture non-invasively in real time.

DETAILED DESCRIPTION:
All subjects will undergo standard management (colposcopy) for their cervical lesion as scheduled. For cervical sites suspicious of dysplasia, acriflavine hydrochloride 0.05% solution will be applied topically, then rinsed with saline prior to in vivo confocal imaging with the hand-held probe. Following that, a biopsy of the suspicious site will be performed irrespective of the confocal microscopy finding. A biopsy of the normal site will be taken for research purposes. The confocal probe imaging will not alter where and how the biopsies will be taken (no change to size of biopsy or location on cervix).

The procedure will add approximately 15 minutes to the duration of the standard outpatient procedure. During each examination, the anatomical location of all tissue areas in question will be recorded using the clock-position nomenclature system. Some normal areas will be also localized and recorded as control. Digital images will be recorded in the computer.

ELIGIBILITY:
Inclusion Criteria:

* indicate understanding of the study
* provide informed consent to participate
* 18 years old or older
* not pregnant and have negative urine pregnancy test
* be schedule for colposcopy & biopsy at the Vancouver General Hospital Women's Clinic

Exclusion Criteria:

* they are breast-feeding
* they had an operation to remove their cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Be scheduled for colposcopy & biopsy at the Vancouver General Hospital Women's Clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Detection of pre-cancer abnormalities of the cervix by the confocal microscopy probe | Probe measurements on participant's cervix should take no more than 10 minutes during the clinical visit

CONTACTS AND LOCATIONS:
Overall Officials: Marette Lee, MD, Principal Investigator — BC Cancer Agency, Gynecologic Oncology
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada